CLINICAL TRIAL: NCT00338949
Title: The Metabolic Syndrome in Patients With Schizophrenia
Brief Title: Ziprasidone for Improving Insulin Sensitivity in People With Schizophrenia Who Are at Risk for Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Pfizer (Industry)
Responsible Party: Principal Investigator, Jonathan M. Meyer, MD, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH074540 (NIH); K23MH074540 (NIH); GA128029 (Other: Pfizer)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia; Metabolic Syndrome X; Insulin Resistance
Keywords: Ziprasidone; Olanzapine; Risperidone; Schizoaffective Disorder; Insulin Sensitivity; Visceral Adiposity; Metabolic Syndrome
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Insulin Resistance; Psychotic Disorders | interventions — ziprasidone; Risperidone; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Participants on risperidone or olanzapine who will remain on risperidone or olanzapine and do not switch to ziprasidone
  Interventions: Drug: Control
- Switch (Experimental): Participants who enter on risperidone or olanzapine and switch to ziprasidone
  Interventions: Drug: Switch

INTERVENTIONS:
Drug: Switch — Participants who are switched to ziprasidone will take a max daily dose of 200 mg, flexibly dosed based on symptoms and adverse effects.
  Other Names: ziprasidone
  Arms: Switch
Drug: Control — Participants will remain taking the same medications of risperidone or olanzapine as they were before study entry.
  Other Names: risperidone; olanzapine
  Arms: Control

SUMMARY:
This study will evaluate the effectiveness of ziprasidone treatment versus treatment with a standard atypical antipsychotic drug in improving insulin sensitivity and reducing excess abdominal fat storage in people with schizophrenia who are at risk for diabetes.

DETAILED DESCRIPTION:
People with schizophrenia often lead more sedentary lifestyles than people without the disease, and they are frequently treated with antipsychotic medications that cause weight gain. Combined, these factors produce an increased risk for metabolic syndrome, which can lead to heart disease and type 2 diabetes. Characteristics of metabolic syndrome include carrying excess weight around the abdominal region; high blood pressure; high blood sugar levels; high levels of fat in the blood; and low levels of HDL cholesterol. Recent studies have shown that certain atypical antipsychotic drugs are relatively weight-neutral. Switching from a drug that promotes weight gain to a weight-neutral medication, such as ziprasidone, may result in significant weight loss. There is insufficient evidence, however, demonstrating the extent of improvement in insulin sensitivity after switching medications. This study will evaluate the effectiveness of ziprasidone treatment versus treatment with a standard atypical antipsychotic drug in improving insulin sensitivity and reducing excess abdominal fat storage in people with schizophrenia who are at risk for diabetes.

Participants in this open label study will currently be undergoing treatment with risperidone or olanzapine at the time of study entry. Upon study entry, they will be randomly assigned to either switch to ziprasidone treatment or remain on their current medications. Both groups will be treated for 26 weeks. Participants will report to the study site for evaluations biweekly until week 10 and then monthly for the duration of the study. The primary outcomes at Week 26 will be: change from baseline in insulin sensitivity, using an intravenous glucose tolerance test; change from baseline in ivisceral fat mass, using a CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Currently receiving antipsychotic therapy with risperidone or olanzapine
* Overweight

Exclusion Criteria:

* Diagnosis of diabetes
* Hospitalization for schizophrenia or schizoaffective disorder within 90 days prior to study entry
* Refractory schizophrenia or schizoaffective disorder
* Currently receiving therapy with clozapine
* No stable residence and phone number for 90 days prior to study entry
* Prior unsuccessful treatment with ziprasidone
* Intolerance to ziprasidone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M. Meyer, MD, Principal Investigator — University of California, San Diego & VA San Diego Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] McEvoy JP, Meyer JM, Goff DC, Nasrallah HA, Davis SM, Sullivan L, Meltzer HY, Hsiao J, Scott Stroup T, Lieberman JA. Prevalence of the metabolic syndrome in patients with schizophrenia: baseline results from the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) schizophrenia trial and comparison with national estimates from NHANES III. Schizophr Res. 2005 Dec 1;80(1):19-32. doi: 10.1016/j.schres.2005.07.014. Epub 2005 Aug 30. PMID 16137860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 06/01/2006. Eligibility: nondiabetic, overweight/obese psychiatrically stable adult outpatients in San Diego with schizophrenia/schizoaffective disorder, on risperidone or olanzapine. Recruitment ended: 12/31/2009
Pre-assignment Details: Exclusions: unstable housing, psychiatric hospitalization in the past 90 days, ongoing substance abuse (except nicotine), history of diabetes mellitus, pregnancy, refractory schizophrenia, prior failure of or intolerance to ziprasidone, oral glucose tolerance test indicative of diabetes mellitus, or corrected QT interval ≥ 500 msec on EKG.
Groups:
- Control: Remain on risperidone or olanzapine.
- Switch: Switch from risperidone or olanzapine to ziprasidone. Ziprasidone will be flexibly dosed based on tolerability and psychiatric response (max dose 200 PO mg/d with food).
Period: Subject Screening
Arm/Group | Control | Switch
Started | 36 | 41
Completed | 25 | 30
Not Completed | 11 | 11
Not completed — Screen failures | 11 | 11
Period: Randomization
Arm/Group | Control | Switch
Started | 25 | 30
Completed | 24 (1 subject withdrew after relapse and hospitalization) | 25 (Reasons for drop out: 2- insomnia 2- symptom exacerbation 1- akathisia)
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 5

BASELINE CHARACTERISTICS:
Population: Nondiabetic, overweight/obese psychiatrically stable adult outpatients with schizophrenia or schizoaffective disorder, on risperidone or olanzapine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Switch | Total
Number analyzed (Participants) | 25 | 30 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.15 (8.15) | 48.73 (8.42) | 48.00 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 19 | 23 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 23 | 26 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 30 | 55
Family Diabetes Mellitus History [Number; unit: participants]
  Family Hx | 4 | 5 | 9
  No Family Hx | 21 | 25 | 46
Smoking Status [Number; unit: participants]
  Smoker | 16 | 18 | 34
  Nonsmoker | 9 | 12 | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.52 (4.49) | 34.64 (7.60) | 33.68 (6.19)
Baseline Antipsychotic [Number; unit: participants]
  Risperidone | 17 | 21 | 38
  Olanzapine | 8 | 9 | 17
PANSS Total Score [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Syndrome Scale Total Score, summed from the positive, negative and general psychopathology subscales. Range 30-210, with higher scores indicating greater psychopathology.
  units on a scale | 62.72 (11.70) | 65.20 (10.66) | 64.07 (11.13)
Central visceral fat volume by CT [Mean (Standard Deviation); unit: mm^3] — Calculated from CT imaging in units of cubic millimeters (mm^3).
  mm^3 | 28442 (10634) | 26939 (12060) | 27622 (11412)
Insulin sensitivity index [Mean (Standard Deviation); unit: (1/mU/L) x 1/Min] — Calculated in units of [(1/(mU/L) x 1/min)]
  (1/mU/L) x 1/Min | 1.596 (1.00) | 1.504 (0.902) | 1.55 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity Index From Baseline to Week 26 ((1/mU/L) x 1/Min)
Description: As measured by frequently sampled intravenous glucose tolerance testing (units: 1/mU/L) x 1/Min)
Time Frame: Measured at Baseline and Week 26
Population: Completers
Measure: Mean (Standard Deviation); unit: (1/mU/L) x 1/Min
Arm/Group | Control | Switch
Number analyzed (Participants) | 24 | 25
(1/mU/L) x 1/Min | 0.072 (0.955) | 0.407 (0.822)
Statistical Analysis 1: Comparison: Control vs Switch; Test type: Superiority or Other; p = 0.228, t-test, 2 sided

2. Primary Outcome: Change in Visceral Fat Mass From Baseline to Week 26
Description: CT measured change in visceral fat mass from baseline to week 26 (mm^3)
Time Frame: Baseline and Week 26
Population: Completers
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Control | Switch
Number analyzed (Participants) | 24 | 25
mm^3 | 315 (5693) | 392 (4340)
Statistical Analysis 1: Comparison: Control vs Switch; Test type: Superiority or Other; p = 0.958, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control | Switch
Serious Adverse Events (participants affected / at risk) | 1/25 | 2/30
Other Adverse Events (participants affected / at risk) | 0/25 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=25) | Switch (N=30)
Psychiatric exacerbation (Psychiatric disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=25) | Switch (N=30)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Akathisia (Psychiatric disorders) | 0 (0) | 1 (1) — Barnes Akathisia Scale

LIMITATIONS AND CAVEATS:
Open label, stable patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No